CLINICAL TRIAL: NCT01341925
Title: Omega-3 Fatty Acids & Psychoeducational Psychotherapy for Childhood Depression
Brief Title: Omega-3 and Therapy Study for Depression
Acronym: OATS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: L. Eugene Arnold (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor-Investigator, L. Eugene Arnold, Principal Investigator, Ohio State University
Organization: Ohio State University (Other)
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2011H0033; 1R34MH085875-01A2 (NIH)
Record Dates: First submitted 2011-04-22; First posted 2011-04-26 (Estimated); Last update posted 2016-03-08 (Estimated); Status verified 2016-03

CONDITIONS: Depression
Keywords: childhood depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Placebo Supplement and No PEP (Placebo Comparator): Will receive two capsules by mouth, two times daily matched for odor and appearance with the active intervention.
  Interventions: Other: Placebo
- Omega-3 and PEP (Experimental): Omega-3 Supplementation will receive 1000 mg Ω3 (two 500 mg capsules, each containing 350 mg EPA: 50 mg DHA; 100 other Ω3)by mouth, two times daily.
  Psychoeducational Psychotherapy (PEP)Therapy sessions occur twice a week for up to 24 sessions of manualized treatment.
  Interventions: Drug: Omega-3 Supplementation; Behavioral: Psychoeducational Psychotherapy (PEP)
- Omega-3 and No PEP (Experimental): Omega-3 Supplementation will receive 1000 mg Ω3 (two 500 mg capsules, each containing 350 mg EPA: 50 mg DHA; 100 other Ω3)by mouth, two times daily.
  Interventions: Drug: Omega-3 Supplementation
- Placebo Supplement and PEP (Experimental): Placebo Supplement will receive two capsules by mouth, two times daily matched for odor and appearance with the active intervention.
  Psychoeducational Psychotherapy (PEP)Therapy sessions occur twice a week for up to 24 sessions of manualized treatment.
  Interventions: Behavioral: Psychoeducational Psychotherapy (PEP)

INTERVENTIONS:
Drug: Omega-3 Supplementation — The Ω3 group will receive 1000 mg Ω3 (two 500 mg capsules, each containing 350 mg EPA: 50 mg DHA; 100 other Ω3) two times daily for a total daily dose of 2000 mg Ω3 (1400 mg EPA: 200 mg DHA; 400 other Ω3). The placebo group will receive two capsules two times daily matched for odor and appearance with the active intervention.
  Other Names: Omega Brite
  Arms: Omega-3 and No PEP; Omega-3 and PEP
Behavioral: Psychoeducational Psychotherapy (PEP) — Therapy sessions occur twice a week for up to 24 sessions of manualized treatment. The importance of separating symptoms from the individual is emphasized. The family is offered support, validation, and recognition for their own difficult experiences in living with the child's mood disorder. Family members are taught that patients are particularly vulnerable to stress and tension; thus, therapists work with families to reduce the level of stress and tension in their homes. Improvement of communication, problem solving and coping strategies can lead to restoration of hope for recovery and decrease family dysfunction. Goals include strengthening the parent-child bond and helping children and parents feel competent to manage depression now and in future recurrences.
  Other Names: IF-PEP
  Arms: Omega-3 and PEP; Placebo Supplement and PEP
Other: Placebo — The placebo group will receive active monitoring (no IF-PEP) and two capsules two times daily matched for odor and appearance with the active intervention.
  Other Names: Pbo
  Arms: Placebo Supplement and No PEP

SUMMARY:
Childhood depression warrants treatment research; including pharmacological and psychotherapeutic interventions. A recent study found fluoxetine to be the only medication with empirical support for decreasing depression in children, but concerns about treatment-emergent suicidal ideation/behavior led the FDA to mandate black-box warning for use of antidepressants in this age group (Bridge et al, 2007). These worries have prompted interest in alternative therapies including dietary supplements such as omega-3 fatty acids (Ω3).

The current study compares Ω3, psychoeducational psychotherapy (PEP), and their combination to a placebo supplement and active monitoring (AM) in a 12-week trial of 60 children with unipolar depression. Primary goals are to determine: 1) feasibility of a) recruiting 60 participants in 24 months; b) retaining participants over a 12-week trial; and 2) effect sizes for Ω3, PEP, and combination treatment. Secondary goals are to explore response curves over time, mediators and moderators, treatment response across an array of outcome variables, adherence to treatment, and side effects. This pilot study of Ω3, PEP, and combined treatment will provide evidence about whether a larger trial is feasible and justifiable.

DETAILED DESCRIPTION:
Approximately 2 to 4% of children experience either major depressive disorder or dysthymic disorder and 5 to 10% of children and adolescents experience subsyndromal depressive symptoms (Birmaher et al). Due to its prevalence and association with significant functioning deficits, childhood depression warrants treatment research. Treatments include pharmacological and psychotherapeutic interventions. A recent meta-analysis found fluoxetine to be the only medication with empirical support for decreasing depression in children, but concerns about treatment-emergent suicidal ideation/behavior led the FDA to mandate black-box warning for use of antidepressants in this age group (Bridge et al, 2007). These worries have prompted interest in alternative therapies including dietary supplements such as omega-3 fatty acids (Ω3). Research on treatment of mood disorders with Ω3 is promising (Schacter et al, 2005); however, only one RCT has been conducted in children, which was positive (Nemets et al, 2006). Findings from other clinical populations (ADHD, adolescent depression, anxiety and pervasive developmental disorders in children) suggest combination treatments are advantageous (Aman et al., 2009; The MTA Cooperative Group, 1999, 2004; The TADS Team, 2007; Walkup et al., 2008). Little is known about the effectiveness of psychotherapy for children age 12 and under who are clinically depressed. Researchers are beginning to develop and test manual-based individual/family therapies for clinic-referred children with diagnosable depression (Kovacs et al, 2006; Tompson et al, 2007); however, no RCTs have been completed. Prior research supports incorporating psychoeducation about depression, support, and skill building to decrease depressive symptoms (Birmaher et al).

The current study compares Ω3, psychoeducational psychotherapy (PEP), and their combination to a placebo supplement and active monitoring (AM) in a 12-week trial of 60 children with unipolar depression. Primary goals are to determine: 1) feasibility of a) recruiting 60 participants in 24 months; b) retaining participants over a 12-week trial; and 2) effect sizes for Ω3, PEP, and combination treatment. Secondary goals are to explore response curves over time, mediators and moderators, treatment response across an array of outcome variables, adherence to treatment, and side effects. This pilot study of Ω3, PEP, and combined treatment will provide evidence about whether a larger trial is feasible and justifiable.

ELIGIBILITY:
Inclusion Criteria:

1. aged 7-14 years (boys and girls)
2. DSM-IV-TR diagnosis of major depressive disorder and/or dysthymic disorder as determined by consensus conference
3. Children's Depression Rating Scale (CDRS-R) score ≥ 40
4. full scale IQ ≥ 70
5. child and at least one parent must be able to complete all assessments
6. child must be able to swallow capsules (training in swallowing will be offered)
7. parent/guardian and child must be willing to have blood drawn from child at two study assessments.

Exclusion Criteria:

1. major medical disorders (eg diabetes, epilepsy, metabolic disorder)
2. inability to communicate in English
3. lack of access via phone
4. autism
5. schizophrenia, or other psychotic states warranting anti-psychotic medication
6. DSM-IV-TR diagnosis of a bipolar disorder
7. active suicidal concern (e.g., "I want to kill myself", a plan for suicide, or an attempt in the past month; however, passive suicidal ideation, such as "I wish I were dead" would not exclude)
8. intake in the previous 4 weeks of supplemental Ω3 fatty acids.

Ages: 7 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 73 (Actual)
Dates: Start 2011-09; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Childhood Depression Rating Scale - Revised (CDRS-R) | Week prior to randomization and then weeks 2, 4, 6, 9, and 12 post-randomization
  The CDRS-R is a severity scale for depression in children ages 6-17. It has 21 items, each rated on a 1-5 or 1-7 point scale in the direction of increasing severity. Scores can range from 17 to 113, demonstrated to correlate significantly with clinical global ratings of depression and to differentiate clinically defined groups of children. Interrater reliability is adequate (r =.86), as is test-retest reliability over a 4 week interval (r =.81; Poznanski et al, 1984). The CDRS-R will be completed at screen to determine clinical impairment of depressive symptoms necessary for study eligibility and at each subsequent assessment to determine clinical response.

SECONDARY OUTCOMES:
K-SADS Depression Rating Scale (KDRS) | Week prior to randomization and then weeks 2, 4, 6, 9, and 12 post-randomization
  Depressive symptom severity for worst past episode(s) and current episode (past two weeks) will be assessed using the KDRS at the assessment visits. The KDRS is a 12-item semi-structured interview with depression symptoms rated on a 6-point scale from none to severe. The KDRS has been shown to be a reliable measure of symptom severity.

CONTACTS AND LOCATIONS:
Overall Officials: L E Arnold, MD, MEd, Principal Investigator — Ohio State University; Mary A Fristad, PhD, Principal Investigator — Ohio State University
Locations (1):
- Ohio State University Medical Center - Harding Hospital, Columbus, Ohio, United States

REFERENCES:
- [Derived] Vesco AT, Young AS, Arnold LE, Fristad MA. Omega-3 supplementation associated with improved parent-rated executive function in youth with mood disorders: secondary analyses of the omega 3 and therapy (OATS) trials. J Child Psychol Psychiatry. 2018 Jun;59(6):628-636. doi: 10.1111/jcpp.12830. Epub 2017 Oct 24. PMID 29063592
- [Derived] Christian LM, Young AS, Mitchell AM, Belury MA, Gracious BL, Arnold LE, Fristad MA. Body weight affects omega-3 polyunsaturated fatty acid (PUFA) accumulation in youth following supplementation in post-hoc analyses of a randomized controlled trial. PLoS One. 2017 Apr 5;12(4):e0173087. doi: 10.1371/journal.pone.0173087. eCollection 2017. PMID 28379964
- [Derived] Young AS, Arnold LE, Wolfson HL, Fristad MA. Psychoeducational Psychotherapy and Omega-3 Supplementation Improve Co-Occurring Behavioral Problems in Youth with Depression: Results from a Pilot RCT. J Abnorm Child Psychol. 2017 Jul;45(5):1025-1037. doi: 10.1007/s10802-016-0203-3. PMID 27604240